CLINICAL TRIAL: NCT06566781
Title: Reinforcement Learning and Obsessive-compulsive Disorder: Exploring the Role of the Orbitofrontal Cortex
Acronym: NEUROCOMP
Status: Recruiting | Type: Observational
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Sponsor
Other Study IDs: NEUROCOMP
Record Dates: First submitted 2024-07-01; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples (30mL: corresponding to 2 tubes EDTA of 6mL each, 2 tubes with clot activator of 6mL each and 1 tube Li+ heparinate of 6mL) from all participants will be collected after clinical assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obsessive-compulsive disorder group: Obsessive-compulsive disorder group: Adult patients (18 to 65 years-old) with obsessive-compulsive (OCD) disorder will be recruited both at Champalimaud Clinical Center and collaborating clinical centers, namely Centro Hospitalar Psiquiátrico de Lisboa, Centro Hospitalar de Lisboa Ocidental and Hospital Garcia de Orta.
- Healthy subjects group: Control subjects group: Adult individuals (18 to 65 years-old) age- and sex-mateched without past or current diagnosis of major neuropsychiatric disorders, including OCD.

SUMMARY:
Obsessive-compulsive disorder (OCD) is a neuropsychiatric condition affecting 1-3% of the population. Typically, symptoms start in adolescence or early adulthood, are time-consuming, and have a significant impact on quality of life. However, first-line approved treatments, based on a combination of pharmacotherapy and psychotherapy, are ineffective in at least 50% of cases. Since the pathophysiology of OCD remains largely unknown, it is expected that a better understanding of the biological mechanisms of OCD would contribute to improved strategies for treatment of the disorder.

Current neurobiological models for OCD highlight the role of corticostriatal dysfunction and hyperactivity of the orbitofrontal cortex (OFC), a part of the prefrontal cortex. Indeed, the lateral OFC plays a crucial role in controlling transitions between automatic, repetitive stimulus-response driven behaviors, and behaviors that reflect the acquisition, by the agent, of a predictive model of the consequences of each action. Previous studies have suggested that the ability to operate this transition is compromised in OCD and may be objectively measured using specifically designed Reinforcement Learning (RL) tasks. Furthermore, growing evidence has suggested that OCD may be associated with systemic immune dysfunction, as has been shown in other common neuropsychiatric conditions, such as depressive disorders. Indeed, there is evidence to support OCD-like symptoms occurring acutely in children after streptococcal infection. These findings have raised the hypothesis that vulnerable individuals exposed to pro-inflammatory early-life environmental risk factors, such as infections and childhood adversity, may suffer neuroinflammatory-induced dysfunction in corticostriatal pathways, increasing the risk of OCD psychopathology.

In this case-control study, the investigators propose an integrative approach to address how structural, functional, and metabolic brain changes involving the corticostriatal circuit correlate with performance in an RL task, as well as with peripheral blood markers of immune dysfunction and associated environmental risk factors such as infection and childhood trauma. Furthermore, since neuromodulation of the prefrontal cortex, using repetitive transcranial magnetic stimulation (rTMS), has recently received FDA clearance for adjunctive treatment in patients with OCD, these associations will be further explored in patients treated with this method. Indeed, in patients with OCD enrolled in the study upon referral to the rTMS Programme for OCD at the Champalimaud Clinical Centre, a follow-up visit will be conducted after the end of treatment (30 sessions of excitatory rTMS over the medial prefrontal cortex). In this subgroup of participants with longitudinal assessment, we will measure change in study parameters and the associations between such change and the clinical effects of treatment, as well as prediction of treatment effects according to baseline assessments.

DETAILED DESCRIPTION:
INTRODUCTION:

Obsessive-compulsive disorder (OCD) is the fourth most common psychiatric disorder, characterized by recurrent and intrusive obsessive thoughts and/or compulsions that are distressing, time-consuming , and a cause of significant impairment. OCD has a lifetime prevalence of 1-3%, and is associated with a reduced life expectancy due to natural and unnatural causes. Current treatments, based on a combination of pharmacotherapy and psychotherapy, are ineffective in at least 50% of cases, with rTMS of the prefrontal cortex having recently received FDA clearance as an adjunctive treatment. Yet, OCD pathophysiology remains largely unknown , and it is expected that a better understanding of OCD 's biological mechanisms would contribute to a better prevention and treatment of the disorder.

Current neurobiological models for the disorder highlight the role of cortico-striatal-thalamo-cortical (CSTC) loops and hyperactivity of the orbitofrontal cortex (OFC), and it has been hypothesized that corticostriatal dysfunction in OCD may occur as an end-consequence of immune and inflammatory dysregulation that leads to structural and functional changes in these circuits. This pathophysiological mechanism was first proposed based on the association between group A β-hemolytic streptococcal (GAS) infection and the abrupt onset of OCD in children, described by Swedo and colleagues (1998) as a distinctive nosologic entity named Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infection (PANDAS). This post-infectious neuropsychiatric syndrome was hypothesized to occur due to a cross-reaction between anti-streptococcal antibodies and the basal ganglia, causing CSTC circuit dysfunction. In addition to GAS, other pathogens have since been suggested as contributing to the development of OCD, albeit no definitive causal associations have been established. Interestingly, childhood adversity, an environmental risk factor for OCD, has also been associated with chronic immune dysfunction in adulthood, namely with increased C-reactive protein, interleukin-6, and tumor necrosis factor (TNF)-α, as well as with increased volume of the right OFC in adult patients with OCD.

While the specific psychopathological consequences of OFC dysfunction in OCD remain unclear, in recent years research in rodents has shown that the OFC, particularly the lateral OFC, is crucial in controlling transitions between automatic, repetitive stimulus-response behaviors (such as habitual behavior in operant-learning tasks, or model-free RL), and behaviors that reflect the acquisition, by the agent, of a predictive model of the consequences of each action (such as goal-directed behavior, or model-based RL). Evidence suggests that patients with OCD may have an abnormal bias towards habitual behavior during operant learning tasks, with subjects having a higher difficulty in developing model-based reinforcement learning strategies. This bias has been proposed to favor the emergence of ritualized compulsive behaviors typical of OCD, and is regarded as a marker of corticostriatal dysfunction that is central to the disorder's pathophysiology.

In this case-control study, the investigators propose an integrative experimental approach to test if structural, functional , and metabolic changes in corticostriatal circuits of patients with OCD correlate with performance in an RL task, as well as with peripheral blood markers of immune dysfunction and early-life environmental risk factors previously implicated in the disorder (e.g., infectious insults and childhood adversities).

STUDY OBJECTIVES:

In this study, the investigators aim to compare patients with OCD and healthy volunteers to assess the association between OCD and:

* Behavioral performance on a RL task;
* Markers of immune dysfunction/autoimmunity in peripheral blood;
* Exposure to proposed environmental risk factors, including infectious agents and childhood adversities;
* Structural and functional brain connectivity patterns, particularly between the OFC and striatum;
* Concentrations of brain metabolites.

The investigators also intend to explore associations of the outcome variables with clinical variables such as obsessive-compulsive symptom severity and age of onset.

Additionally, for patients enrolled in this study who will undergo rTMS for clinical purposes at our clinical center, the investigators aim to assess if there is an association between the behavioral, neuroimaging, and immunological variables and treatment response. Specifically, the investigators will test 1) if post-treatment changes in behavioral and neuroimaging measures correlate with treatment response, and 2) if baseline behavioral, neuroimaging, and immune measures predict response to treatment. Specifically, the investigators will test:

* if rTMS treatment will alter performance in the RL task and if such changes correlate with response to treatment;
* if rTMS modulates organizational patterns in large-scale neural networks and in the functional and structural connectivity between OFC and striatum, and if these changes correlate with response to treatment or to changes in performance of the RL task;
* if rTMS leads to changes in metabolite concentrations in the OFC and striatum and if these are associated with response to treatment or with changes in performance of the RL task;
* if environmental risk factors and baseline peripheral markers of immune dysfunction, brain structural and functional connectivity correlates, and baseline concentration of metabolites in the OFC and striatum predict the outcome of rTMS both in terms of OCD symptom change and in terms of RL task performance.

PROCEDURES:

For this study, the investigators will recruit 115 age- and sex-matched subjects with OCD and 115 control volunteers. After signing informed consents, participants will complete a thorough clinical assessment, including confirmation of psychiatric diagnoses using the appropriate modules of the Structured Clinical Interview for DSM-5, and rating of obsessive-compulsive symptoms using the Yale-Brown Obsessive-Compulsive Scale II, the gold-standard structured clinical interview for OCD assessment. Other clinical variables of interest will be assessed using the following instruments:

* Mini International Neuropsychiatric Interview (M.I.N.I.) - Portuguese or English version. The version used for this study does not include the module for Psychopathy.
* Yale-Brown Obsessive-Compulsive Scale-II - Portuguese or English version
* State-Trait Anxiety Inventory - Portuguese or English version
* Beck Depression Inventory-II - Portuguese or English version
* Childhood Trauma Questionnaire - Portuguese or English version
* Perceived Stress Scale - Portuguese or English version
* Barratt Impulsiveness Scale - Portuguese or English version
* Edinburgh Handedness Inventory - Portuguese or English version After completing the clinical assessment, participants will proceed to blood collection for measurement of peripheral blood markers of immune dysfunction/autoimmunity. This will be followed by performance of a RL task on a computer, and lastly by a magnetic resonance imaging session. The protocol for the latter will comprise a T1 sequence for structural assessment, resting-state BOLD images (rs-fMRI) of the whole brain, Diffusion Weighted Imaging (DWI) to measure diffusivity of water molecules within the brain, and brain tissue concentration of metabolites using Magnetic Resonance Spectroscopy (MRS) analysis of two voxels, one in the left OFC and the other in the left caudate.

For the subgroup of patients enrolled in the study that will undergo rTMS for clinical purposes at our Champalimaud Clinical Programme, the investigators will propose a follow-up visit after completion of the treatment. In this visit, participants will be asked to repeat the clinical assessment, RL task , and the MRI protocol as described before. The clinical TMS protocol comprises 30 sessions of excitatory rTMS (20 Hz) over the medial prefrontal cortex, as defined by international guidelines, using a protocol that includes individualized symptom provocation before each stimulation session, to elicit a moderate level of obsessional distress, as reported by patients. This subgroup will also complete all the procedures of experiment 1 prior to initiating the rTMS treatment protocol. After the last session of rTMS treatment, up to one week after the treatment has ended, these participants will repeat the RL task and the MRI protocol as described for baseline.

DATA COLLECTION:

* Clinical assessment: Clinical interview and psychometric instruments (self-report questionnaires and semi-structured interviews);
* Behavioral assessment: Participants will perform a RL task in the form of a computer game;
* Blood sample collection: A blood sample will be collected, processed on the same day, and stored in a -80ºC freezer;
* MRI protocol: MRI sequences will be acquired on a 3T Phillips scanner with a 32-channel head coil. The imaging protocol will include T1-weighted sequence using a 3-dimensional fast field echo (FFE); resting-state BOLD echo-planar imaging (EPI); DTI EPI sequence with b values of 0, 1000 , and 2000 s/mm2. For each b value, 64 equally spaced gradient directions will be sampled. Magnetic Resonance Spectroscopy (MRS) with a Point-Resolved Spectroscopy (MEGA-PRESS) pulse sequence will be used to acquire signals from hydrogen protons to measure spectra from metabolites in the OFC and striatum. The total scan time will be around 50 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Exclusively for the OCD group: established diagnosis of Obsessive-Compulsive Disorder according to DSM-5 criteria;
* Exclusively for the control group: does not meet DSM criteria for any of the psychiatric diagnoses screened by the Mini International Neuropsychiatric Interview;
* Age between 18 and 65 years-old;
* Fluent Portuguese or English speaker.

Exclusion Criteria:

* Any acute medical illness;
* Substance abuse or dependence;
* Pregnancy;
* Dementia;
* Developmental disorders with low intelligence quotient or any other form of cognitive impairment;
* Active neurological disease;
* Previously known structural lesion of the central nervous system;
* Illiteracy or otherwise not understanding the study's instructions;
* Inability to give informed consent;
* Individuals presenting with any psychotic or mood disorder condition requiring hospitalization at that moment;
* For experiment 2, these exclusion criteria will be expanded by additional factors that specifically preclude TMS use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be adults, aged 18 to 65 years, that will be recruited either for the clinical or control group. The clinical population will include individuals with OCD diagnosis, according to the following inclusion criteria. The two groups will be matched by age and sex.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of high sensitivity C Reactive Protein (hsCRP). | Baseline.
  Serum concentration of hsCRP, expressed in mg/dL, as measured by enzyme-linked immunosorbent assay (ELISA).
Seropositivity for Group A Streptococcus (GAS). | Baseline.
  Number of participants who are seropositive for GAS measured by anti-streptolysin O (ASO) antibodies (IgG).
Basal ganglia and orbito-frontal cortex (OFC) volume. | Baseline.
  Volume of basal ganglia structures (e.g. caudate, putamen and globus pallidus) and the OFC, in cubic milimeters.
Exposure to childhood trauma as measured by the Childhood Trauma Questionnaire (CTQ). | Baseline.
  Exposure to childhood trauma measured by the CTQ. The total score varies between 25 and 125, providing an overall measure of the exposure to childhood trauma, with higher scores representing exposure to more (and more severe) traumatic events.
Obsessive-compulsive symptom severity. | Baseline and longitudinal (up to one week after finishing rTMS treatment protocol).
  Obsessive-compulsive symptom severity as measured by Yale-Brown Obsessive-Compulsive Scale II (YBOCS-II). YBOCS-II total score ranges between 0 and 50, with higher scores relating to higher severity of obsessive-compulsive symptoms.
Measurement of fractional anisotropy (FA) in the brain white matter. | Baseline and longitudinal (up to one week after finishing rTMS treatment protocol).
  Voxel-wise FA measures obtained from diffusion-weighted imaging (DWI).
Functional connectivity of the orbitofrontal cortex (OFC). | Baseline and longitudinal (up to one week after finishing rTMS treatment protocol).
  Voxel-wise FA measures obtained from diffusion-weighted imaging (DWI).
Concentration of N-acetyl-aspartate (NAA) and N-acetyl-aspartyl-glutamate (NAAG). | Baseline and longitudinal (up to one week after finishing rTMS treatment protocol).
  Concentration of NAA and NAAG measured by Magnetic Resonance Spectroscopy (MRS) in the left caudate and left subcortical OFC, expressed in mmol/L.
Model-free component in a computational model of a reinforcement learning behavioral task. | Baseline and longitudinal (up to one week after finishing rTMS treatment protocol).
  Weight of the model-free component in a computational model of behavior where behavior is assumed to be controlled by a weighted sum of model-based and model-free components.

SECONDARY OUTCOMES:
Peripheral concentration of cytokines. | Baseline
  Plasmatic concentration of cytokines (interferon gamma (IFN-γ), tumor necrosis factor (TNF-α), interleukin (IL)-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, IL-17 and IL-23), expressed In pg/mL, as measured by ELISA.
Peripheral concentration of transforming growth factor (TGF)-β. | Baseline
  Plasmatic concentration of TGF-β, expressed in pM, as measured by ELISA.
Presence of auto-antibodies. | Baseline
  Number of participants positive for auto-antibodies such as anti-basal ganglia (ABGA), anti-nuclear (ANA), and anti-thyroid antibodies.
Seropositivity for Toxoplasma gondii, Cytomegalovirus (CMV), Herpes simplex virus (HSV1 and HSV2). | Baseline
  Number of participants who are seropositive for IgG Toxoplasma gondii, CMV, HSV1 and HSV2 antibodies.
Measurement of Neurite Orientation Dispersion and Density Imaging (NODDI) in the brain white matter. | Baseline and longitudinal (up to one week after finishing rTMS treatment protocol).
  Voxel-wise NODDI measures obtained from diffusion-weighted imaging (DWI).

OTHER OUTCOMES:
Gene expression of peripheral cytokines. | Baseline
  Genetic expression of peripheral cytokines (IFN-γ, TNF-α, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12, IL-17, IL-23 and TGF-β), expressed in cycle thresholds (CT), as measured by quantitative Real-Time Polymerase Chain Reaction (RT-PCR).
Functional connectivity pattern supported in lesional OCD neuroanatomy. | Baseline
  Voxel-wise functional connectivity of the regions-of-interest extracted from lesional network mapping analyses of cases with secondary OCD.
Measurement of Mean Kurtosis (MK) in the brain white matter. | Baseline
  Voxel-wise MK obtained from DWI.

CONTACTS AND LOCATIONS:
Overall Officials: Albino J Oliveira-Maia, MD MPH PhD, Principal Investigator — Director of Neuropsychiatry, Champalimaud Research & Clinical Centre, Champalimaud Foundation
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AMERICAN PSYCHIATRIC ASSOCIATION. Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Diagnostic and Statistical Manual of Mental Disorders 4th edition TR 2013;:280.
- [Background] Sasson Y, Zohar J, Chopra M, Lustig M, Iancu I, Hendler T. Epidemiology of obsessive-compulsive disorder: a world view. J Clin Psychiatry. 1997;58 Suppl 12:7-10. PMID 9393390
- [Background] CALDAS DE ALMEIDA J, XAVIER M, CARDOSO G et al. Estudo Epidemiológico Nacional de Saúde Mental - 1.o Relatório. Lisboa Faculdade de Ciências Médicas, da 2013;:60.
- [Background] Hollander E, Bienstock CA, Koran LM, Pallanti S, Marazziti D, Rasmussen SA, Ravizza L, Benkelfat C, Saxena S, Greenberg BD, Sasson Y, Zohar J. Refractory obsessive-compulsive disorder: state-of-the-art treatment. J Clin Psychiatry. 2002;63 Suppl 6:20-9. PMID 12027116
- [Background] Carmi L, Alyagon U, Barnea-Ygael N, Zohar J, Dar R, Zangen A. Clinical and electrophysiological outcomes of deep TMS over the medial prefrontal and anterior cingulate cortices in OCD patients. Brain Stimul. 2018 Jan-Feb;11(1):158-165. doi: 10.1016/j.brs.2017.09.004. Epub 2017 Sep 6. PMID 28927961
- [Background] Ruffini C, Locatelli M, Lucca A, Benedetti F, Insacco C, Smeraldi E. Augmentation effect of repetitive transcranial magnetic stimulation over the orbitofrontal cortex in drug-resistant obsessive-compulsive disorder patients: a controlled investigation. Prim Care Companion J Clin Psychiatry. 2009;11(5):226-30. doi: 10.4088/PCC.08m00663. PMID 19956460
- [Background] Nauczyciel C, Le Jeune F, Naudet F, Douabin S, Esquevin A, Verin M, Dondaine T, Robert G, Drapier D, Millet B. Repetitive transcranial magnetic stimulation over the orbitofrontal cortex for obsessive-compulsive disorder: a double-blind, crossover study. Transl Psychiatry. 2014 Sep 9;4(9):e436. doi: 10.1038/tp.2014.62. PMID 25203167
- [Background] Saxena S, Rauch SL. Functional neuroimaging and the neuroanatomy of obsessive-compulsive disorder. Psychiatr Clin North Am. 2000 Sep;23(3):563-86. doi: 10.1016/s0193-953x(05)70181-7. PMID 10986728
- [Background] Milad MR, Rauch SL. Obsessive-compulsive disorder: beyond segregated cortico-striatal pathways. Trends Cogn Sci. 2012 Jan;16(1):43-51. doi: 10.1016/j.tics.2011.11.003. Epub 2011 Dec 2. PMID 22138231
- [Background] Pauls DL, Abramovitch A, Rauch SL, Geller DA. Obsessive-compulsive disorder: an integrative genetic and neurobiological perspective. Nat Rev Neurosci. 2014 Jun;15(6):410-24. doi: 10.1038/nrn3746. PMID 24840803
- [Background] Gray SM, Bloch MH. Systematic review of proinflammatory cytokines in obsessive-compulsive disorder. Curr Psychiatry Rep. 2012 Jun;14(3):220-8. doi: 10.1007/s11920-012-0272-0. PMID 22477442
- [Background] Pearlman DM, Vora HS, Marquis BG, Najjar S, Dudley LA. Anti-basal ganglia antibodies in primary obsessive-compulsive disorder: systematic review and meta-analysis. Br J Psychiatry. 2014 Jul;205(1):8-16. doi: 10.1192/bjp.bp.113.137018. PMID 24986387
- [Background] Menzies L, Chamberlain SR, Laird AR, Thelen SM, Sahakian BJ, Bullmore ET. Integrating evidence from neuroimaging and neuropsychological studies of obsessive-compulsive disorder: the orbitofronto-striatal model revisited. Neurosci Biobehav Rev. 2008;32(3):525-49. doi: 10.1016/j.neubiorev.2007.09.005. Epub 2007 Oct 17. PMID 18061263
- [Background] Balleine BW, O'Doherty JP. Human and rodent homologies in action control: corticostriatal determinants of goal-directed and habitual action. Neuropsychopharmacology. 2010 Jan;35(1):48-69. doi: 10.1038/npp.2009.131. PMID 19776734
- [Background] Yin HH, Knowlton BJ, Balleine BW. Lesions of dorsolateral striatum preserve outcome expectancy but disrupt habit formation in instrumental learning. Eur J Neurosci. 2004 Jan;19(1):181-9. doi: 10.1111/j.1460-9568.2004.03095.x. PMID 14750976
- [Background] Yin HH, Ostlund SB, Knowlton BJ, Balleine BW. The role of the dorsomedial striatum in instrumental conditioning. Eur J Neurosci. 2005 Jul;22(2):513-23. doi: 10.1111/j.1460-9568.2005.04218.x. PMID 16045504
- [Background] Gremel CM, Costa RM. Orbitofrontal and striatal circuits dynamically encode the shift between goal-directed and habitual actions. Nat Commun. 2013;4:2264. doi: 10.1038/ncomms3264. PMID 23921250
- [Background] Gillan CM, Papmeyer M, Morein-Zamir S, Sahakian BJ, Fineberg NA, Robbins TW, de Wit S. Disruption in the balance between goal-directed behavior and habit learning in obsessive-compulsive disorder. Am J Psychiatry. 2011 Jul;168(7):718-26. doi: 10.1176/appi.ajp.2011.10071062. Epub 2011 May 15. PMID 21572165
- [Background] SUTTON RS, BARTO AG. Introduction to Reinforcement Learning. Learning 1998;4:1-5.
- [Background] Dolan RJ, Dayan P. Goals and habits in the brain. Neuron. 2013 Oct 16;80(2):312-25. doi: 10.1016/j.neuron.2013.09.007. PMID 24139036
- [Background] Daw ND, Niv Y, Dayan P. Uncertainty-based competition between prefrontal and dorsolateral striatal systems for behavioral control. Nat Neurosci. 2005 Dec;8(12):1704-11. doi: 10.1038/nn1560. Epub 2005 Nov 6. PMID 16286932
- [Background] Voon V, Derbyshire K, Ruck C, Irvine MA, Worbe Y, Enander J, Schreiber LR, Gillan C, Fineberg NA, Sahakian BJ, Robbins TW, Harrison NA, Wood J, Daw ND, Dayan P, Grant JE, Bullmore ET. Disorders of compulsivity: a common bias towards learning habits. Mol Psychiatry. 2015 Mar;20(3):345-52. doi: 10.1038/mp.2014.44. Epub 2014 May 20. PMID 24840709
- [Background] Attwells S, Setiawan E, Wilson AA, Rusjan PM, Mizrahi R, Miler L, Xu C, Richter MA, Kahn A, Kish SJ, Houle S, Ravindran L, Meyer JH. Inflammation in the Neurocircuitry of Obsessive-Compulsive Disorder. JAMA Psychiatry. 2017 Aug 1;74(8):833-840. doi: 10.1001/jamapsychiatry.2017.1567. PMID 28636705
- [Background] Williams KA, Swedo SE. Post-infectious autoimmune disorders: Sydenham's chorea, PANDAS and beyond. Brain Res. 2015 Aug 18;1617:144-54. doi: 10.1016/j.brainres.2014.09.071. Epub 2014 Oct 7. PMID 25301689
- [Background] Orlovska S, Vestergaard CH, Bech BH, Nordentoft M, Vestergaard M, Benros ME. Association of Streptococcal Throat Infection With Mental Disorders: Testing Key Aspects of the PANDAS Hypothesis in a Nationwide Study. JAMA Psychiatry. 2017 Jul 1;74(7):740-746. doi: 10.1001/jamapsychiatry.2017.0995. PMID 28538981
- [Background] Sutterland AL, Fond G, Kuin A, Koeter MW, Lutter R, van Gool T, Yolken R, Szoke A, Leboyer M, de Haan L. Beyond the association. Toxoplasma gondii in schizophrenia, bipolar disorder, and addiction: systematic review and meta-analysis. Acta Psychiatr Scand. 2015 Sep;132(3):161-79. doi: 10.1111/acps.12423. Epub 2015 Apr 15. PMID 25877655
- [Background] Keenan KE, Ainslie M, Barker AJ, Boss MA, Cecil KM, Charles C, Chenevert TL, Clarke L, Evelhoch JL, Finn P, Gembris D, Gunter JL, Hill DLG, Jack CR Jr, Jackson EF, Liu G, Russek SE, Sharma SD, Steckner M, Stupic KF, Trzasko JD, Yuan C, Zheng J. Quantitative magnetic resonance imaging phantoms: A review and the need for a system phantom. Magn Reson Med. 2018 Jan;79(1):48-61. doi: 10.1002/mrm.26982. Epub 2017 Oct 30. PMID 29083101
- [Background] Reichenbach JR, Venkatesan R, Schillinger DJ, Kido DK, Haacke EM. Small vessels in the human brain: MR venography with deoxyhemoglobin as an intrinsic contrast agent. Radiology. 1997 Jul;204(1):272-7. doi: 10.1148/radiology.204.1.9205259.
- [Background] Desmond JE, Glover GH. Estimating sample size in functional MRI (fMRI) neuroimaging studies: statistical power analyses. J Neurosci Methods. 2002 Aug 30;118(2):115-28. doi: 10.1016/s0165-0270(02)00121-8. PMID 12204303
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Machii K, Cohen D, Ramos-Estebanez C, Pascual-Leone A. Safety of rTMS to non-motor cortical areas in healthy participants and patients. Clin Neurophysiol. 2006 Feb;117(2):455-71. doi: 10.1016/j.clinph.2005.10.014. Epub 2006 Jan 4. PMID 16387549
- [Background] Schrader LM, Stern JM, Koski L, Nuwer MR, Engel J Jr. Seizure incidence during single- and paired-pulse transcranial magnetic stimulation (TMS) in individuals with epilepsy. Clin Neurophysiol. 2004 Dec;115(12):2728-37. doi: 10.1016/j.clinph.2004.06.018. PMID 15546781
- [Background] Jahanshahi M, Ridding MC, Limousin P, Profice P, Fogel W, Dressler D, Fuller R, Brown RG, Brown P, Rothwell JC. Rapid rate transcranial magnetic stimulation--a safety study. Electroencephalogr Clin Neurophysiol. 1997 Dec;105(6):422-9. doi: 10.1016/s0924-980x(97)00057-x. PMID 9448643
- [Background] Kim DR, Epperson N, Pare E, Gonzalez JM, Parry S, Thase ME, Cristancho P, Sammel MD, O'Reardon JP. An open label pilot study of transcranial magnetic stimulation for pregnant women with major depressive disorder. J Womens Health (Larchmt). 2011 Feb;20(2):255-61. doi: 10.1089/jwh.2010.2353. PMID 21314450